CLINICAL TRIAL: NCT05673512
Title: To Evaluate IAH0968 in Combination With CAPEOX in a Phase II/III Clinical Study of HER2-positive Metastatic Colorectal Cancer
Brief Title: To Evaluate IAH0968 in Combination With CAPEOX in HER2-positive Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: SUNHO（China）BioPharmaceutical CO., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IAH0968-202
Record Dates: First submitted 2023-01-03; First posted 2023-01-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: HER2 Gene Mutation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IAH0968+ CAPEOX (Active Comparator): IAH0968+ CAPEOX in HER2 positive metastatic colorectal cancer patient
  Interventions: Combination Product: Injection of IAH0968 + CAPEOX
- CAPEOX (Active Comparator): PLACEBO+CAPEOX in HER2 positive metastatic colorectal cancer patient
  Interventions: Combination Product: PLACEBO+CAPEOX

INTERVENTIONS:
Combination Product: Injection of IAH0968 + CAPEOX — PLACEBO+CAPEOX in HER2 positive metastatic colorectal cancer patient
  Arms: IAH0968+ CAPEOX
Combination Product: PLACEBO+CAPEOX — PLACEBO+CAPEOX in HER2 positive metastatic colorectal cancer patient
  Arms: CAPEOX

SUMMARY:
The Phase IIa of this clinical study, a dose-escalation study of IAH0968 in combination with CAPEOX, is designed for safety and tolerability in subjects with HER2-positive advanced or metastatic solid tumors. Phase IIb/III is an operational seamless adaptive design consisting of two phases. Phase I (Phase IIb) was designed to initially evaluate the efficacy and safety of IAH0968+CAPEOX in HER2-positive subjects with metastatic colorectal cancer, using PFS.

DETAILED DESCRIPTION:
The Phase IIa of this clinical study, a dose-escalation study of IAH0968 in combination with CAPEOX regimen, was designed to evaluate Safety and tolerability of IAH0968+CAPEOX regimen in subjects with HER2-positive advanced or metastatic solid tumors.

Phase IIb/III uses an operational seamless adaptive design and consists of two phases. Phase I (Phase IIb) aims to initially evaluate the efficacy and safety of IAH0968+CAPEOX in HER2-positive subjects with metastatic colorectal cancer by PFS. Phase II (Phase III) was designed to evaluate the efficacy and safety of IAH0968+CAPEOX versus placebo +CAPEOX in HER2-positive subjects with metastatic colorectal cancer using PFS.

ELIGIBILITY:
Inclusion criteria:

1. Stage IIa only: advanced or metastatic solid tumor confirmed by histopathology or cytology.
2. Only stage IIb and III: Patients with mCRC confirmed by histopathology or cytology, who are not suitable for radical surgical excision or local therapy, and who have not previously received systemic antitumor therapy for CRC (including systemic chemotherapy, molecular targeted drug therapy, biotherapy and investigational therapy, and have completed adjuvant chemotherapy for ≥6 months) can be admitted to the group.
3. Age range from 18 to 75 years old (including the critical value), gender is not limited.
4. Proof of HER2-positive (IHC) 3+, or IHC 2+ and FISH +, by immunohistochemical (IHC) staining and/or fluorescence in situ hybridization (FISH), and wild type KRAS, NRAS, and BRAF genes. HER2 positive status was interpreted according to the current Chinese guidelines for detecting HER2 in gastric cancer.
5. According to the researchers' judgment, CAPEOX scheme is suitable.
6. At least one measurable lesion according to RECIST 1.1 criteria (tumor lesion located in the area of prior radiotherapy or other local regional treatment site is generally not considered as a measurable lesion unless it shows definite progression or persists three months after radiotherapy).
7. The physical status score of the Eastern Oncology Consortium (ECOG) was 0-1.
8. Expected survival ≥3 months.
9. Adequate organ function: 1) Blood system (no blood transfusion or hematopoietic stimulating factor treatment within 14 days) : absolute neutrophil count (ANC) ≥1.5×109/L, platelet count (PLT) ≥90×109/L, hemoglobin (HGB) ≥90 g /L; Liver function: total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN), except for Gilbert syndrome; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3.0 times ULN, liver metastasis or liver cancer patients need AST and ALT≤5.0 times ULN. 3. Renal function: serum creatinine (Cr) ≤1.5 ULN; If creatinine Creatinine clearance (Ccr) ≥50 ml/min (calculated by Cockcroft-Gault formula) was required at 1.5 ULN. Coagulation function: prothrombin International Normalized ratio (INR) ≤1.5 ULN, activated partial thrombin time (APTT) ≤1.5 ULN.
10. Eligible patients (male and female) who are fertile must agree to use a reliable contraceptive method (hormonal or barrier method or abstinence) with their partner during the trial period and for at least 6 months after the last medication; Women of reproductive age must have a negative blood or urine pregnancy test 7 days before first use of the study drug.
11. Subjects must give informed consent to the study prior to the study and voluntarily sign written informed consent.

Exclusion criteria:

1. Stage IIa only: chemotherapy, radiotherapy, biotherapy, endocrine therapy, immunotherapy and other antitumor therapies were received within 4 weeks prior to the first use of the study drug, except for the following: 1 nitrosourea or mitomycin C was used within 6 weeks prior to the first use of the study drug; 2 Oral administration of fluoripyritics and small molecule targeted drugs 2 weeks prior to the first use of the study drug or within 5 half-lives of the drug, whichever is longer; 3 Chinese patent drugs with anti-tumor indications were used within 2 weeks prior to the first use of the investigational drug.
2. Have received other investigational drugs or treatments that are not on the market within 4 weeks prior to use of the investigational drug.
3. Stage IIa only: Adverse reactions to previous antitumor therapy have not yet returned to the NCI CTCAE 5.0 scale evaluation ≤ Level 1 or relevant provisions of inclusion criteria (except for toxicities without safety risks as determined by the investigators, such as alopecia, grade 2 peripheral neurotoxicity, stable hypothyroidism after hormone replacement therapy, etc.).
4. Known hypersensitivity to any antibody-class drug (NCI CTCAE 5.0 rating ≥3) or to investigational drug, CAPEOX protocol active ingredient or inactive excipients.
5. Confirmed mismatch repair defect (dMMR) or high microsatellite instability (MSI-H) solid tumors (unless subject is unable to receive immune checkpoint inhibitors due to a pre-existing medical condition, or unknown MSI/MMR status).
6. Had major organ surgery (excluding needle biopsy) or significant trauma, or required elective surgery, within 4 weeks prior to initial use of the study drug.
7. Received systemic administration of corticosteroids (prednisone > 10 mg/day or equivalent dose of the same drug) or other immunosuppressant therapy, except: treatment with topical, ocular, intraarticular, intranasal, and inhaled corticosteroids; Short-term use of glucocorticoids for prophylactic treatment (e.g. to prevent shadow allergy).
8. Use of immunomodulatory drugs within 14 days (Appendix 5).
9. Received any live vaccine within 4 weeks prior to the first administration of the study drug.
10. Have previously received allogeneic hematopoietic stem cell transplantation or organ transplantation.
11. There are clinical symptoms of brain parenchymal metastasis or meningeal metastasis. Patients with BMS who had been treated were enrolled if magnetic resonance imaging (MRI) or computed tomography (CT) showed no signs of progression at least 8 weeks after the end of treatment and 4 weeks before the first use of the study drug.
12. There is an active infection that currently requires intravenous anti-infective therapy.
13. A history of immunodeficiency, including a positive test for human immunodeficiency virus (HIV) antibodies.
14. Active hepatitis B (HBsAg positive and HBV-DNA≥1.0×103 copies /mL or ≥2000IU/mL, active hepatitis C (HCV-RNA> 1.0×103 copies /mL or > 100 IU/mL).
15. Severe and uncontrollable lung disease (severe infectious pneumonia, interstitial lung disease, etc.).
16. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to: 1. Have serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmias requiring clinical intervention, degree II-III atrioventricular block, etc.; 2 QT interval (QTcF) mean corrected by Fridericia method > 470 ms;3 Acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or above cardiovascular and cerebrovascular events occurred within 6 months prior to initial administration;4 Present with heart failure or left ventricular ejection fraction (LVEF)&lt of the New York Heart Association (NYHA) cardiac function grade ≥II; 50%;5. Clinically uncontrollable hypertension.
17. Have an active or past autoimmune disease with a risk of recurrence (e.g., systemic lupus erythematosus, class Rheumatoid arthritis, vasculitis), clinically stable autoimmune thyroid disease, type I diabetes, vitiligo, Children with cured atopic dermatitis and psoriasis that does not require systemic treatment (within the last 2 years) are excluded.
18. Non-melanoma skin cancer that has been clinically cured for more than 2 years and is currently suffering from other malignant tumors, limitations Exceptions include prostate cancer, carcinoma in situ (such as cervical carcinoma in situ), etc.
19. There was clinically uncontrollable third space effusion, which was not suitable for inclusion by the investigator.
20. Known alcohol or drug dependence.
21. Have mental disorders or poor compliance.
22. Pregnant or lactating women.
23. The investigator believes that the subjects have a history of other serious systemic diseases or are not suitable to participate in this clinical study for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival（PFS） | 12 months
  treatment index

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No